CLINICAL TRIAL: NCT04606628
Title: OPTIEgg- Optimal Value Increase of Egg Products
Brief Title: Optimal Value Increase of Egg Products
Acronym: OPTIEgg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Nofima (Other); Norwegian University of Life Sciences (Other); Nortuna (Unknown); Norilia (Unknown); Orkla (Unknown); Danægg (Unknown)
Responsible Party: Principal Investigator, Stine Marie Ulven, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020/95084/REK Sør-Øst
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy; Inflammation; Aging
Keywords: Eggshell membrane; Healthy volunteers; Old volunteers
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This study is a randomized double-blinded controlled trial and is considered as a pilot study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One of the employees will distribute the capsules and know which of the group is placebo and intervention. Everyone else involved in the project will be blinded for this knowledge.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will consume 2 capsules containing eggshell membrane(ESM) with breakfast every day in 4 weeks.
  Interventions: Other: Eggshell membrane (ESM)
- Placebo (Experimental): Participants will consume 2 capsules with no bioactive substance (placebo) with breakfast every day in 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Eggshell membrane (ESM) — The intervention group will consume two capsules containing (in total) 500mg ESM with breakfast every day in 4 weeks.
  Arms: Intervention
Other: Placebo — The placebo group will consume two placebo capsules (Cellulose) with breakfast every day in 4 weeks
  Arms: Placebo

SUMMARY:
The aim of this project is to evaluate daily intake of eggshell membrane taken as supplement (capsule), will reduce markers of inflammation in older people.

ELIGIBILITY:
Inclusion Criteria:

The study will include home-dwelling men and women ≥ 70 years. All subjects have to be in a good enough condition to meet up at the Department of Nutrition, University of Oslo at two occasions during the study period.

Exclusion Criteria:

* CRP >10 mg/L
* Egg allergy
* Use of medication affecting inflammation
* Unstable use of medication or supplements last 3 months
* Unwilling to keep the physical activity level, habitual dietary intake, tobacco use and weight stable during the study period
* Severe illness last 3 months
* Unwilling to perform physical tests
* Eligibility
* Diabetes type I or II, HbA1c ≥ 6.5 %

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in plasma levels of inflammatory markers | Measured at baseline and after 4 weeks (end of study)
  concentration of C-reactive protein (CRP)
Change in plasma levels of inflammatory markers | Measured at baseline and after 4 weeks (end of study)
  concentration of TNFalpha

SECONDARY OUTCOMES:
Changes in body composition - measured by Bioimpedance (BIA) | Measured at baseline and after 4 weeks
  fat free mass (% and kg), fatt mass (% and in kg)
Change in muscle strength | Measured at baseline and after 4 weeks
  Measured by grip strength
Changes in markers related to lipid metabolism | Measured at baseline and after 4 weeks
  Blood concentrations of e.g. triglycerides, total-, LDL- and HDL- cholesterol, free fatty acids and lipoprotein subclasses
Peripheral blood mononuclear cell (PBMC) gene expression | Measured at baseline and after 4 weeks
  mRNA levels of of genes involved in lipid metabolism and inflammation
Change in microbiota composition (optional) | Measured at baseline and after 4 weeks
  Consenctration of faecal short-chain fatty acids
Change in microbiota composition (optional) | Measured at baseline and after 4 weeks
  bacteria type and diversity
Changes in satiety hormones | Measured at baseline and after 4 weeks
  e.g. concentration of serum ghrelin, amylin, leptin
Changes in metabolome plasma profile | Measured at baseline and after 4 weeks
  concentration of amino acids in blood
Changes in metabolome plasma profile | Measured at baseline and after 4 weeks
  concentration of low molecular molecules in blood
Changes in body weight | Measured at baseline and after 4 weeks
  Weight (kg) measured by digital scale
Changes in body mass index (BMI) | Measured at baseline and after 4 weeks
  Measured as body weight in kg/height in meter2 ( kg/m2)
Changes in physical performance | Measured at baseline and after 4 weeks
  Short Physical Performance Battery (SPPB) test (includes balance test, chair test (sit to stand) and walk test)

CONTACTS AND LOCATIONS:
Overall Officials: Stine M Ulven, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway